CLINICAL TRIAL: NCT01291771
Title: Detection and Outcomes of Myocardial Microvascular Disease in Patients With End Stage Renal Disease
Brief Title: Myocardial Microvascular Disease in ESRD
Acronym: MICROCARD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2010.611
Record Dates: First submitted 2011-02-07; First posted 2011-02-08 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: End Stage Renal Disease; Myocardial Microvascular Disease
Keywords: End stage renal disease; myocardial microvascular disease; cardiorenal syndrome; coronary flow reserve; index of microvascular resistance; Patients with end stage renal disease scheduled or not for kidney or kidney + pancreatic transplantation
MeSH Terms: conditions — Kidney Failure, Chronic; Cardio-Renal Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- comparator (Other): One group of patients with no myocardial ischemia on non invasive testing will be followed up for 2 years
  Interventions: Procedure: Invasive FFR + CFR measurements are performed during coronary angiography using a pressure guide wire
- coronary angiography group (Experimental): One group of patients with myocardial ischemia on non invasive testing will undergo coronary angiography and measure of FFR + CFR to detect myocardial microvascular disease
  Interventions: Procedure: Invasive FFR + CFR measurements are performed during coronary angiography using a pressure guide wire

INTERVENTIONS:
Procedure: Invasive FFR + CFR measurements are performed during coronary angiography using a pressure guide wire — The guide is placed in the distal segment of the coronary artery to measure instantaneously distal pressure and temperature with a tip sensor. Proximal pressure and temperature are being measured from the probe used to catheterize the coronary vessel and from the shaft of the guide. After basal measurement, intracoronary injection of 150µg of adenosine is performed to induce peripheral vasodilatation leading to hyperaemia in the vessel. Additional injection of 3mL 0.9% saline bolus at room temperature at the time of hyperaemia is performed to calculate CFR from transit mean time. FFR and CFR are being recorded at the time of hyperaemia. Subsequently IMR is being calculated from distal pressure and transit mean time. The measurements will be performed in the LAD, circumflex and right coronary arteries.

SUMMARY:
Cardiovascular diseases are the leading cause of mortality in patients with end stage renal disease (ESRD). They often have myocardial ischemia (a major predictor of mortality) on non invasive testing (Stress echocardiography and/or myocardial perfusion scintigraphy) but the incidence of significant coronary stenosis (>70%) is low. The goal of this observational study is to evaluate the incidence and clinical outcomes of proven myocardial microvascular disease in patients with end stage renal disease scheduled or not for kidney transplantation. These patients routinely undergo non invasive detection of myocardial ischemia. Patient included in the study will be followed up for 2 years for major cardiovascular events. Patients with detected myocardial ischemia during non invasive testing are being explored by coronary angiography. During coronary angiography additional detection of myocardial microvascular disease is being performed by simultaneous measurement of Fractional Flow Reserve (FFR) and Coronary Flow Reserve (CFR) followed by calculation of the index of microcirculatory resistance (IMR).

Comparison of cardiovascular outcomes between patients with and without myocardial ischemia and patients with and without myocardial microvascular disease will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients age > 18 years with end stage renal disease under dialysis and/or scheduled for kidney or kidney + pancreatic transplantation
* Having a non invasive detection of myocardial ischemia and agreeing to participate (signed informed consent document)

Exclusion Criteria:

Past medical history of

* Acute coronary syndrome
* Hypertrophic cardiomyopathy
* severe aortic and/or mitral valvular disease (grade ≥ 3)
* Known contraindications to adenosine injection: AV block grade ≥ 2 and/or sinoatrial block unless prior implantation of a pace maker, asthma, allergic reaction to adenosine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-01; Primary Completion 2014-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Major cardiovascular events | Inclusion: 1 year - Follow up: 2 years
  Major cardiovascular events
  * Death (all cause)
  * Acute coronary syndromes (STEMI, NSTEMI, UA)
  * New onset of stable angina
  * New onset of congestive heart failure or progression of previously known congestive heart failure (need for therapeutic intensification and/or hospital admission)
  * Cardiogenic shock
  * Stroke
  * Severe cardiac arrhythmia (FV, VT)
  * New onset of atrial fibrillation

SECONDARY OUTCOMES:
Incidence of myocardial microvascular disease detected by FFR + CFR in ESRD patients with myocardial ischemia on non invasive tests. | Inclusion: 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Denis ANGOULVANT, Dr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Service de Cardiologie D - Hôpital Louis Pradel - Hospices Civils de Lyon, Bron, France

REFERENCES:
- [Derived] Bejan-Angoulvant T, Bergerot C, Juillard L, Mezergues A, Morelon E, Pouteil-Noble C, Andre-Fouet X, Angoulvant D. Myocardial microvascular disease and major adverse cardiovascular events in patients with end-stage renal disease: rationale and design of the MICROCARD study. Nephrol Dial Transplant. 2012 Jul;27(7):2886-91. doi: 10.1093/ndt/gfs008. Epub 2012 Feb 17. PMID 22344775